CLINICAL TRIAL: NCT02710864
Title: A Cross-sectional Study of Congenital Cytomegalovirus Infection in Newborns in China
Status: Completed | Type: Observational
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Vice dean of School of Public Health,Xiamen University, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: CMV-EPI-003
Record Dates: First submitted 2016-03-05; First posted 2016-03-17 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples With DNA — saliva and urine samples of the newborns
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of this study were to evaluate the incidence of congenital CMV infection in neonates, and assess the concordance of detecting congenital cytomegalovirus (CMV) infection in neonatal saliva and urine samples.

DETAILED DESCRIPTION:
This Cross-sectional study was conducted to recruit neonates less than 14 days old delivered in Maternal and Child Health Hospitals (MCHHs) of Xinmi City, Jiaxian County, Zhongmu County and Huli District Xiamen City, in China, from June 2015 to June 2016. The aim of this study is to enroll ~1800 neonates, and collect their saliva and urine samples which will be tested the CMV DNA by using real-time PCR.

ELIGIBILITY:
Inclusion Criteria:

* Neonates aged 0 to 14 days
* Neonates delivered in MCHHs of Xinmi City, Jiaxian County, Zhongmu County and Huli District Xiamen City

Exclusion Criteria:

* the parents of neonates not comply with our study

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates aged 0 to 14 days in MCHHs of Xinmi City, Jiaxian County, Zhongmu County and Huli District Xiamen City, in China ,were recruited, after written informed consents provided by the parents.
Sampling Method: Probability Sample
Enrollment: 1510 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of cCMV infection in newborns | up to 5 months

SECONDARY OUTCOMES:
the Kappa value of CMV prevalence between saliva and urine samples | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Professor, Principal Investigator — Xiamen University
Locations (4):
- China (4):
  - Maternity and Child care of Huli District, Xiamen, Fujian
  - Maternity and Child care of Jiaxian County, Pingdingshan, Henan
  - Maternity and Child care of Xinmi City, Zhengzhou, Henan
  - Maternity and Child care of Zhongmu County, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided